CLINICAL TRIAL: NCT05018949
Title: Evaluation of Post-Angioplasty Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2021-08-22; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have undergone LL angioplasty: Patients who have undergone LL angioplasty are enrolled in study for a medical records review.
  Interventions: Procedure: Lower limb angioplasty

INTERVENTIONS:
Procedure: Lower limb angioplasty — Patients who have undergone LL angioplasty are enrolled in study for a medical records review.

SUMMARY:
There is no hard and fast rule guiding the clinical decision between angioplasty and amputation. As such, this decision is greatly dependant on each clinician's experience and preference as to whether treatment should be conservative or aggressive.

Angioplasty can help restore blood flow and long-term patency of the blood vessels can help prevent major surgeries, such as amputation which affects patient's quality of life. However, some of these patients do not benefit from angioplasty and eventually had to undergo amputation. On the other hand, there are patients that undergo amputation, but may stand to benefit from angioplasty. Hence, it is essential to identify patients that will likely benefit from angioplasty to increase limb salvage rate. Many studies performed have also concluded that before amputations are performed, surgeons should consider angioplasty procedures.

Through a medical record review of patients that have undergone angioplasty to evaluate post-angioplasty outcomes, we hope to identify factors that potentially affects these outcomes. Ultimately with a better understanding of these factors and their impact on angioplasty outcomes, a predictive model or guideline can be developed to identify patients that stands to benefit from angioplasty. Such a model can help clinicians to better counsel patients on the risk and benefits, alternatives and prognosis. Patients can also make a better informed decision regarding their treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted into SGH Department of Vascular Surgery, and have successfully undergone angioplasty

Exclusion Criteria:

* Minors under age of 21

Ages: 21 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients that have successfully undergone lower limb angioplasty procedures
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Amputation Free Survival | 12 months post-op
  Freedom from major limb amputation
Freedom from target lesion revascularization | 12 months post-op
  Freedom from any interventions to the index treated lesion
Primary Patency | 12 months
  Patency of the treated lesion at index procedure
Wound healing rates | 12 months
  Healing of index wounds and whether there is any recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No